CLINICAL TRIAL: NCT03919695
Title: Development and Pilot Testing of a Combination Intervention to Reduce Heavy Drinking and Improve HIV Care Engagement Among Fisherfolk in Uganda
Brief Title: Development of an Intervention to Reduce Heavy Drinking and Improve HIV Care Engagement Among Fisherfolk in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Makerere University (Other); Mildmay Uganda Limited (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R34AA025891 (NIH); R34AA025891 (NIH)
Record Dates: First submitted 2019-04-07; First posted 2019-04-18 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; HIV-infection/Aids
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome | interventions — Mass Screening; Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kisoboka: structural and behavioral intervention (Experimental): The KISOBOKA intervention adapts and combines a behavioral intervention with a structural component. The behavioral intervention component includes, alcohol screening, financial literacy training, and counseling and goal setting related to savings, alcohol use, and HIV care engagement. The structural intervention component changes the mode of work payment from cash to mobile money.
  Interventions: Behavioral: Kisoboka: Behavioral and Structural Intervention
- Screening and Referral (Active Comparator): Brief feedback on AUDIT-C score, referral for alcohol counseling, and briefly discussion of the importance of HIV care engagement and adherence.
  Interventions: Behavioral: Screening and Referral

INTERVENTIONS:
Behavioral: Kisoboka: Behavioral and Structural Intervention — The intervention has two components; a structural component and a behavioral component. The intervention draws from behavioral economics and motivational interviewing.
  Structural component: This component is about receiving work payments via mobile money instead of cash.
  Behavioral component: This component includes feedback on alcohol screening, counseling, client-centered goal setting, self-monitoring, financial literacy training, and text message reminders of life/savings and healthy living goals.
  Other Names: KISOBOKA
  Arms: Kisoboka: structural and behavioral intervention
Behavioral: Screening and Referral — Alcohol screening and referral and emphasizing the importance of HIV care engagement and ART adherence
  Arms: Screening and Referral

SUMMARY:
Fisherfolk are a high risk population for HIV and are prioritized to receive antiretroviral treatment (ART) in Uganda, but risky alcohol use among fisherfolk is a barrier to HIV care engagement; multilevel factors influence alcohol use and poor access to HIV care in fishing villages, including a lack of motivation, social support, access to savings accounts, and access to HIV clinics. This project aims to address these barriers, and subsequently reduce heavy alcohol use and increase engagement in HIV care, through an intervention in which counselors provide individual and group counseling to increase motivation, while also addressing structural barriers to care through increased opportunities for savings and increased social support. This may be a feasible approach to help this hard-to-reach population reduce drinking and increase access care, which could ultimately reduce mortality rates, improve treatment outcomes, and through its effect on HIV viral load, decrease the likelihood of transmitting HIV to others.

DETAILED DESCRIPTION:
The investigators propose to develop and pilot a brief combination intervention which addresses the key drivers of alcohol use and barriers to HIV care engagement and ART adherence in this population. This study addresses these multi-level factors in an intervention which combines a structural component of changing the mode of work payments from cash to mobile money, to reduce "cash in the pocket," and increase the accessibility of savings through mobile phone-based banking services, with behavioral components to change behavior. For the behavioral components, the study combines and adapt two efficacious Motivational Interviewing (MI)-based alcohol interventions to the cultural and situational context of this population: a brief intervention tested in Kenya and an intervention rooted in behavioral economics which focuses on increasing the extent to which individuals' behavior is motivated by and consistent with their long-term goals such as saving money for the future-in which the structural component of the intervention is interwoven. The aims of the project are to: 1) Combine a promising structural (e.g., reducing "cash in the pocket") and behavioral intervention to promote reductions in heavy alcohol use, engagement in HIV care, and ART adherence among HIV+ male fisherfolk. These interventions will be adapted and tailored to the population to create the proposed KISOBOKA ("It is possible!") intervention. The investigators will refine the combination intervention through qualitative research with HIV+ male fisherfolk and community stakeholders and an initial pilot test with 15 participants examining acceptability and feasibility; 2) Pilot the intervention, randomizing to the KISOBOKA intervention arm (n=80) or to the control arm (n=80, alcohol screening and referral). The investigators will assess feasibility, acceptability, and preliminary estimates of the potential for the intervention, as compared to control, to decrease heavy drinking frequency and improve HIV care engagement and ART adherence through 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* occupation of working in the fishing industry or industry supporting the fishing industry; HIV+; on ART for at least 1 month; missed one or more dose of ART in the prior 2 weeks; consume 5 or more drinks per occasion 2 or more times in the prior month or have an AUDIT-C score of 4 or greater; not planning to move from the area within the next 6 weeks; have their own mobile phone and can be reached via phone

Exclusion Criteria:

* currently receiving a majority of income for work via mobile money, does not speak Luganda or English, unable to read basic Luganda or English, occupation of boat or engine owner.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Kiene, Principal Investigator — San Diego State University
Locations (1):
- selected Wakiso District HIV clinics, Multiple Locations, Wakiso District, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from HIV clinics and enrolled in the trial between January 2021 and March 2022.
Groups:
- Structural and Behavioral Intervention: The KISOBOKA intervention adapts and combines a behavioral intervention with a structural component. The behavioral intervention component includes, alcohol screening, financial literacy training, and counseling and goal setting related to savings, alcohol use, and HIV care engagement. The structural intervention component changes the mode of work payment from cash to mobile money.
  Behavioral and Structural Intervention: The intervention has two components; a structural component and a behavioral component. The intervention draws from behavioral economics and motivational interviewing.
  Structural component: This component is about receiving work payments via mobile money instead of cash.
  Behavioral component: This component includes feedback on alcohol screening, counseling, client-centered goal setting, self-monitoring, financial literacy training, and text message reminders of life/savings and healthy living goals.
- Screening and Referral: Brief feedback on AUDIT-C score, referral for alcohol counseling, and briefly discussion of the importance of HIV care engagement and adherence.
  Screening and Referral: Alcohol screening and referral
Period: 3-month Follow-up
Arm/Group | Structural and Behavioral Intervention | Screening and Referral
Started | 80 | 80
Completed | 79 | 75
Not Completed | 1 | 5
Not completed — Death | 1 | 1
Not completed — unable to contact | 0 | 3
Not completed — in prison | 0 | 1
Period: 6-month Follow-up
Arm/Group | Structural and Behavioral Intervention | Screening and Referral
Started (All participants not deceased at 3-months were attempted to be followed-up at 6 months since some at 3-months were unreachable due to being imprisoned or having traveled far away. As shown in the next flow (completed any follow-up) 2 participants in the screening and referral arm who were "lost" at 3 months completed the 6-month follow-up and contribute to longitudinal analyses.) | 79 | 79 (Participants not deceased (those who were in prison or were unable to be contacted at 3-months) were attempted to be followed up for the 6 month follow-up)
Completed | 78 | 74
Not Completed | 1 | 5
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — in prison | 0 | 2
Period: Any Follow-up (3 and/or 6 Month)
Arm/Group | Structural and Behavioral Intervention | Screening and Referral
Started (This flow illustrates analyses using baseline, 3 month, and 6 month data. For these analyses participants having baseline and at least one follow-up are included. Therefore, this aspect of the flow represents participants with (baseline and) 3 and/or 6 month follow-up completed.) | 80 (This period represents participants who started the study at baseline (80) and completed any follow-up (3 or 6-month) and were thus included in analyses of outcomes assessed at both follow-up time points.) | 80 (This period represents participants who started the study at baseline (80) and completed any follow-up (3 or 6-month) and were thus included in analyses of outcomes assessed at both follow-up time points.)
Completed | 79 | 77
Not Completed | 1 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Structural and Behavioral Intervention | Screening and Referral | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.26 (6.29) | 39.01 (6.70) | 38.14 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 80 | 80 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 80 | 80 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 80 | 80 | 160
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 80 | 80 | 160
Occupation [Count of Participants; unit: Participants]
  Fishing | 51 | 50 | 101
  Other | 29 | 30 | 59
Education [Count of Participants; unit: Participants]
  Greater than grade 7 | 18 | 24 | 42
  Grade 7 or less | 62 | 56 | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hazardous Alcohol Use at Baseline, 3 and 6 Month Follow up
Description: hazardous alcohol use as assessed with the Alcohol Use Disorders Identification Test - Concise (AUDIT-C) measure using a cutpoint of 9 to indicate hazardous alcohol use in this population
Time Frame: 3 and 6 month follow up
Population: Participants completing baseline and at least one follow-up are included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Kisoboka: Structural and Behavioral Intervention: The KISOBOKA intervention adapts and combines a behavioral intervention with a structural component. The behavioral intervention component includes, alcohol screening, financial literacy training, and counseling and goal setting related to savings, alcohol use, and HIV care engagement. The structural intervention component changes the mode of work payment from cash to mobile money.
  Kisoboka: Behavioral and Structural Intervention: The intervention has two components; a structural component and a behavioral component. The intervention draws from behavioral economics and motivational interviewing.
  Structural component: This component is about receiving work payments via mobile money instead of cash.
  Behavioral component: This component includes feedback on alcohol screening, counseling, client-centered goal setting, self-monitoring, financial literacy training, and text message reminders of life/savings and healthy living goals.
Arm/Group | Kisoboka: Structural and Behavioral Intervention | Screening and Referral
Number analyzed (Participants) | 79 | 77
Participants
  Baseline, AUDIT-C greater than/equal to 9 | 41 | 26
  3-month follow-up, AUDIT-C greater than/equal to 9: number analyzed (Participants) | 79 | 75
  3-month follow-up, AUDIT-C greater than/equal to 9 | 18 | 27
  6-month follow-up, AUDIT-C greater than/equal to 9: number analyzed (Participants) | 78 | 74
  6-month follow-up, AUDIT-C greater than/equal to 9 | 15 | 20
Statistical Analysis 1: Comparison: Screening and Referral; Generalized Estimating Equations (GEE) model specifying a logistic distribution examining the time x arm interaction; Test type: Superiority; p = .002, GEE model specifying a logistic distribu; Odds Ratio (OR) = .29, 95% CI 2-sided [.11 to .73] — time x arm effect for the comparison at 6-month follow-up

2. Primary Outcome: Change in Phosphatidylethanol (PEth) From Baseline
Description: alcohol biomarker which correlates well with the volume of alcohol consumed over the prior 2-4 weeks
Time Frame: 6 month follow up
Population: Participants who completed the 6-month follow-up
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kisoboka: Structural and Behavioral Intervention | Screening and Referral
Number analyzed (Participants) | 78 | 74
ng/mL
  baseline | 554.30 (607.15) | 518.34 (521.77)
  6-month follow-up | 479.95 (459.63) | 595.65 (656.93)

3. Primary Outcome: Number of Participants With Optimal Antiretroviral (ART) Adherence at Baseline, 3 and 6 Month Follow up
Description: Adult AIDS Clinical Trials Group (AACTG) measure. Self-reported ART adherence for the past 4 days. Optimal adherence >=90%.
Time Frame: 3 and 6 month follow up
Population: Participants completing baseline and at least one follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Structural and Behavioral Intervention | Screening and Referral
Number analyzed (Participants) | 79 | 77
Participants
  baseline | 55 | 57
  3-months: number analyzed (Participants) | 79 | 75
  3-months | 55 | 40
  6-months: number analyzed (Participants) | 78 | 74
  6-months | 49 | 37

4. Secondary Outcome: Change From Baseline in Frequency of Consuming ≥ 5 Drinks/Occasion in the Prior 28 Days
Description: number of days consumed ≥ 5 standard drinks/occasion in the 28 days prior to the assessment. 1 drink = 10g pure alcohol. Self-reported
Time Frame: 3 and 6 month follow up
Population: Participants completing baseline and at least one follow-up assessment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kisoboka: Structural and Behavioral Intervention | Screening and Referral
Number analyzed (Participants) | 79 | 77
days
  baseline | 7.77 (6.31) | 8.45 (7.47)
  3 months: number analyzed (Participants) | 79 | 75
  3 months | 6.87 (6.81) | 8.52 (7.63)
  6 months: number analyzed (Participants) | 78 | 74
  6 months | 7.85 (7.25) | 8.46 (7.52)

5. Secondary Outcome: Number of Participants With an HIV Viral Load Value <839 at Baseline and Follow-up, From Clinic Records Viral Load Tests for Routine Clinical Monitoring
Description: The proportion of participants with an HIV viral load test value of <839 using clinical data among those with viral load tests available. Viral load tests were PCR-based assays. These clinics used a value of <839 to indicate a suppressed HIV viral load. The use of clinic records data relied on participants having routine viral load tests at intervals corresponding to the measurement intervals of baseline or before and near follow-up. Baseline: sample taken before baseline (up to 294 days before) and follow-up includes samples taken between 126-330 days after baseline.
Time Frame: approximately 6 month follow up
Population: Participants with a routine clinic viral load assessment taken within one of the study measurement time windows (baseline or follow-up) - thus a participant with a viral load test recorded in the clinic record at either time point is included. It is expected that not all participants contribute data for this outcome nor have data at both time points. A participant is included if they have data at either time point, resulting in a larger overall number analyzed than the number at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Kisoboka: Structural and Behavioral Intervention | Screening and Referral
Number analyzed (Participants) | 63 | 59
Participants
  baseline HIV viral load <839 (from clinic records): number analyzed (Participants) | 56 | 55
  baseline HIV viral load <839 (from clinic records) | 42 | 44
  follow-up HIV viral load <839 (from clinic records): number analyzed (Participants) | 29 | 24
  follow-up HIV viral load <839 (from clinic records) | 24 | 18

6. Secondary Outcome: HIV Care Engagement
Description: missed visit count, visit adherence, 3 month visit constancy
Time Frame: 6 month follow up
Reporting Status: Not Posted, anticipated posting 2025-06

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Structural and Behavioral Intervention | Screening and Referral
All-Cause Mortality (participants affected / at risk) | 1/80 | 2/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03919695/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03919695/ICF_001.pdf